CLINICAL TRIAL: NCT05624723
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics, Safety, and Pharmacodynamics of INCB054707 in Participants With Normal and Impaired Renal Function and Participants on Hemodialysis
Brief Title: Study to Evaluate the Pharmacokinetics, Safety, and Pharmacodynamics of INCB054707 in Participants With Normal and Impaired Renal Function and Participants on Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB054707-106; NCT05694195 (obsolete NCT alias)
Record Dates: First submitted 2022-11-11; First posted 2022-11-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Renal Insufficiency; Kidney Diseases
Keywords: renal impairment; hemodialysis; Kidney failure; end-stage renal disease
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Normal Renal Function (Experimental): Participants with normal levels of renal function will receive a single oral dose of INCB054707 75 mg on Day 1.
  Interventions: Drug: INCB054707
- Group 2: Mild Renal Impairment (Experimental): Participants with mild levels of renal function will receive a single oral dose of INCB054707 75 mg on Day 1.
  Interventions: Drug: INCB054707
- Group 3: Moderate Renal Impairment (Experimental): Participants with moderate levels of renal function will receive a single oral dose of INCB054707 75 mg on Day 1.
  Interventions: Drug: INCB054707
- Group 4: Severe Renal Impairment (Experimental): Participants with severe levels of renal function will receive a single oral dose of INCB054707 75 mg on Day 1.
  Interventions: Drug: INCB054707
- Group 5: Kidney Failure (Experimental): Group 5 participants with ESRD maintained on HD will receive a single dose of INCB054707 across 2 treatment periods before (Period 1) and after (Period 2) an HD session in order to study the effects of HD on INCB054707.
  Interventions: Drug: INCB054707

INTERVENTIONS:
Drug: INCB054707 — INCB054707 75 mg will be administered orally
  Other Names: Povorcitinib

SUMMARY:
This is a multi-center, open-label, parallel-group study to evaluate oral doses of INCB054707 in participants with varying levels of renal function or impairment.

ELIGIBILITY:
Inclusion Criteria:

* Classification at screening by renal function based on eGFR as calculated by the MDRD formula and requirement for HD (Group 5).
* Participants eligible for Group 5 with ESRD have received HD for at least 3 months prior to screening.
* Participants eligible for Group 1 should be in good health as determined by no clinically significant deviations from normal for medical history, physical examination, vital signs, 12-lead ECGs, or clinical laboratory determinations at screening or Day -1.
* Participants eligible for Groups 2 through 5 may have medical findings consistent with their degree of renal dysfunction, as determined by medical history, physical examination, vital signs, 12-lead ECGs, and clinical laboratory determinations at screening and Day -1 (Groups 2 through 4) or Period 1 Day -1 (Group 5).
* Body mass index within the range of 18.0 to 40.0 kg/m2 (inclusive) at screening.
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, hepatic, GI, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening or evidence of rapidly deteriorating renal function.
* Current, functioning organ transplant or a cheduled organ transplant within 6 weeks after check-in.
* History of malignancy within 5 years of screening, with the exception of cured basal cell carcinoma, squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* History of clinically significant GI disease or surgery (cholecystectomy and appendectomy are allowed) that could impact the absorption of study drug.
* Eligible for Group 1 and have a history of renal disease or renal injury as indicated by an abnormal, clinically significant renal function profile at screening or Day -1.
* Eligible for Groups 2 through 5 and have had a change in disease status within 30 days of screening, as documented by the participant's medical history and deemed clinically significant by the investigator.
* History or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study, including any of the following:

  1. Recent myocardial infarction (within 6 months of check-in)
  2. New York Heart Association Class III or IV congestive heart failure
  3. Unstable angina (within 6 months of check-in)
  4. Clinically significant (symptomatic) cardiac arrhythmias (eg, sustained ventricular tachycardia, second- or third-degree atrioventricular block without a pacemaker)
  5. Uncontrolled hypertension
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank within 4 weeks of screening (within 2 weeks for plasma only).
* Blood transfusion within 4 weeks of Day -1 (for Groups 1 through 4) or Period 1 Day -1 (Group 5).
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment.
* Positive test and symptomatic for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization for or immunity due to infection with HBV may be included at the discretion of the investigator.
* Eligible for Group 1 and have a history of using tobacco- or nicotine-containing products within 6 months of screening.
* Eligible for Groups 2 through 5 and smoke > 10 cigarettes per day or equivalent use of other tobacco- or nicotine-containing products and are unwilling to refrain from tobacco or nicotine use on dosing days and abide by CRU restrictions.
* History of alcohol dependency within 3 months of screening.
* Positive breath test for ethanol or positive urine or saliva screen for drugs of abuse (confirmed by repeat test) at screening or check-in that are not otherwise explained by permitted concomitant medications.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) of study drug administration with another investigational medication or current enrollment in another investigational drug study.
* Current treatment or treatment within 15 days or 5 half-lives (whichever is longer) before the first dose of study drug with moderate and potent inducers or inhibitors of CYP3A4 (refer to the Drug Interaction Database Program [University of Washington School of Pharmacy 2002] for prohibited drugs).
* Consumption of Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices within 72 hours before the first dose of study drug.
* Eligible for Group 1 and have used prescription drugs within 14 days of study drug administration or nonprescription medications/products (including vitamins, minerals, and hytotherapeutic/herbal/plant-derived preparations) within 7 days of study drug administration. However, occasional use of acetaminophen and ibuprofen is permitted (see Section 6.6.1).
* Eligible for Groups 2 through 5 and have used prescription drugs within 14 days of study drug administration, with the exception of established therapy for renal disease and the treatment of associated disorders that have been stable for at least 7 days prior to study drug administration, as approved by the investigator and in consultation with the sponsor's medical monitor.
* Current or recent history (within 30 days before screening) of a clinically significant bacterial, fungal, parasitic, or mycobacterial infection, currently receiving systemic antibiotics, or having a current clinically significant viral infection at screening or check-in.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Inability to undergo venipuncture or tolerate venous access.
* Eligible for Group 5 and not expected to continue HD treatment for the duration of the study.
* Women who are pregnant or breastfeeding.
* Use of hormonal contraception
* QTcF > 450 milliseconds for Groups 1 through 3 and QTcF > 470 milliseconds for Group 4.
* Eligible for Group 1 and have abnormal LFT values, defined as aspartate aminotransferase, alanine aminotransferase, and serum (total and direct) bilirubin, as well as amylase and lipase above the upper limit of the normal range at screening.
* Eligible for Groups 2 through 4 and have values outside the normal ranges for LFTs; however, values may be acceptable if they are consistent with the participant's renal condition (if stable for 1 month prior to screening) and if the investigator (or designee) and the sponsor feel that the results are not clinically significant (based on age and renal impairment status).
* Receipt of live (including attenuated) vaccines within 3 months of check-in or anticipation of need for such a vaccine during the study (Note: Nonlive or inactivated vaccines are allowed up to 2 weeks prior to the first dose of study drug).
* Known hypersensitivity or severe reaction to INCB054707 or excipients of INCB054707 (refer to the IB).

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Parameter: Cmax of INCB054707 | Days 1-4
  Defined as maximum observed plasma concentration of INCB054707
Pharmacokinetics Parameter: AUC0-t of INCB054707 | Days 1-4
  Area Under the concentration- time curve up to the last measurable concentration of INCB054707
Pharmacokinetics Parameter: AUC0-∞ of INCB54707 | Days 1-4
  Defined as under the concentration-time curve up to the last measurable concentration of INCB054707

SECONDARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAE'S) | Up to 21 days
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Pharmacokinetics Parameter: tmax of INCB054707 | Days 1-4
  Defined as time to reach maximum plasma concentration of INCB054707; during dialysis for Group 5 Period 1.
Pharmacokinetics Parameter: t½ of INCB054707 | Days 1-4
  Defined as apparent terminal-phase disposition half-life of INCB054707; during dialysis for Group 5 Period 1.
Pharmacokinetics Parameter: CL/F of INCB054707 | Days 1-4
  Defined as oral dose clearance of INCB054707; during dialysis for Group 5 Period 1.
Pharmacokinetics Parameter: Vz/F of INCB054707 | Days 1-4
  Defined as apparent oral dose volume of distribution; during dialysis for Group 5 Period 1.
Pharmacokinetics Parameter: AUC3-7 of INCB054707 | Days 1-4
  Defined as area under the concentration-time curve from 1 to 5 of INCB054707; during dialysis for Group 5 Period 1.

CONTACTS AND LOCATIONS:
Locations (2):
- Orlando Clinical Research Center, Orlando, Florida, United States
- Apex Gmbh, Munich, Germany

IPD SHARING:
Plan to Share IPD: No